CLINICAL TRIAL: NCT05851131
Title: Surveying Knowledge, Attitudes, and Practices of Primary Care Physicians in Turkey Regarding Osteoporosis Management.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: AHek1
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family physicians: Family physicians working in Turkey who gave consent to participate in the study.
  Interventions: Other: Approach to Diagnosis and Treatment of Osteoporosis Questionnaire

INTERVENTIONS:
Other: Approach to Diagnosis and Treatment of Osteoporosis Questionnaire — The survey will use multiple-choice questions to assess primary care physicians' knowledge on the diagnosis and treatment of osteoporosis. The questions will cover various aspects, including medication options, their mechanisms of action, side effects, and recommended vitamin D supplementation dosages. The physicians will also be asked about their sources of knowledge and how they keep themselves updated on the topic, as well as their self-evaluation of their knowledge. Background information, such as their professional and demographic characteristics, will also be collected. The survey questionnaire used in other studies will be adapted for this survey based on the "Updated approach for the management of osteoporosis in Turkey: a consensus report."

SUMMARY:
This study aims to assess the knowledge of primary care physicians on the diagnosis and treatment of osteoporosis.

DETAILED DESCRIPTION:
Multiple choice questions will be used to assess information related to the diagnosis and treatment of osteoporosis, including knowledge of various medications, their mechanisms of action and side effects, and recommended dosage of vitamin D supplementation. The participating physicians will also be asked about their sources of knowledge acquisition and how they keep updated on this topic, as well as their self-evaluation of knowledge. Furthermore, background information will be collected, including professional and demographic characteristics. A questionnaire previously used in other studies will be adapted for the study based on the 'Updated approach for the management of osteoporosis in Turkey: a consensus report'.

ELIGIBILITY:
Inclusion Criteria:

* Giving consent.
* Working as a family physician assistant, family physician specialist or general practitioner in Turkey.

Exclusion Criteria:

* Not giving consent.
* Having any physical or mental illness that may prevent reading, understanding and filling out the form.

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Family physician assistants, family physician specialists and general practitioners working in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge levels, attitudes and practices of primary care physicians in Turkey | 1 day
  The survey will use multiple-choice questions to assess primary care physicians' knowledge on the diagnosis and treatment of osteoporosis. The questions will cover various aspects, including medication options, their mechanisms of action, side effects, and recommended vitamin D supplementation dosages. The physicians will also be asked about their sources of knowledge and how they keep themselves updated on the topic, as well as their self-evaluation of their knowledge. Background information, such as their professional and demographic characteristics, will also be collected. The survey questionnaire used in other studies will be adapted for this survey based on the "Updated approach for the management of osteoporosis in Turkey: a consensus report."

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request by the corresponding author.